CLINICAL TRIAL: NCT00491595
Title: Phase I Multiple-Dose Clinical Study of Soy Isoflavones in Healthy, Post-Menopausal Women
Brief Title: Phase I Clinical Study of Soy Isoflavones in Healthy, Post-Menopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: NCI-N01-CN-75035
Expanded Access: Available
Record Dates: First submitted 2007-06-22; First posted 2007-06-26 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-06

CONDITIONS: Drug Toxicity
Keywords: Soy isoflavones; Genotoxicity; Apoptosis; Estrogenic effects
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Soybean Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: High Dose Soy isoflavones

SUMMARY:
The purpose of this research study is to examine the safety of specific soy components, known as isoflavones, and to find out what effects (good and bad) these components have on tissues that are sensitive to the hormone estrogen in healthy, post-menopausal women. Isoflavones are compounds that occur naturally in soybeans and can be extracted to put in to capsule form or add to foods. The capsule formulation being used in this study is considered an investigational drug. This research is being done because many scientists believe that isoflavones may play a role in the prevention of some kinds of cancer. While isoflavones have been safely consumed in foods for centuries, we need to know if these soy components are safe to take in higher doses when they are extracted from foods and provided in a supplement form. We plan to test the safety and effects of the soy isoflavones known as genistein, daidzein and glycitein.

DETAILED DESCRIPTION:
This will be a double blind, Phase I, multiple dose clinical trial of orally administered soy isoflavones (PTI G-2535, 70% unconjugated isoflavones containing genistein, daidzein, and glycitein). This preparation will be referred to as soy isoflavones in this and all study related documents to more accurately reflect the study drug's content. The multiple dose trial will last four months (112 days) and will include healthy, post-menopausal women as determined by FSH levels and lack of spontaneous bleeding for at least one year. After eligibility is determined, all potential subjects will ingest a soy shake to determine if they are producers of the daidzein metabolite, equol. We expect to find approximately 30% of our eligible subjects to be equol-producers as published in the literature. Equol producers will be defined as individuals with plasma levels >20ug/L; non-equol producers as those with <10ug/L 37. Individuals with intermediate equol values (> 10 ug/L to < 20 ug/L) will be excluded from the study. Stratified randomization will assign the subjects to one of the two groups, aiming for 30-40% equol producers in each group. Group 1 (20 subjects) will receive a dietary supplement containing 600 mg of genistein in two doses of 300 mg (as part of a soy isoflavones mixture) per day orally administered over an 84-day period. Group 2 (10 subjects) will receive a placebo supplement (excipients from the active formulation), orally administered over an 84-day period. These women will be recruited from the local population within the Research Triangle area. The study will be conducted at the UNC Hospital General Clinical Research Center (GCRC).

ELIGIBILITY:
Inclusion Criteria:

* Performance status 0, 1, or 2 on ECOG scale
* Acceptable hematopoietic, hepatic, and renal function (WBC≥3500 µL, platelet count ≥ 100,000/ml, serum creatinine < 2.0 mg/dl, serum bilirubin ≤ 2.0 mg/dl, transaminases < two times normal limits)
* Post-menopausal status - FSH level > 27 mIU/ml, no spontaneous bleeding > 1 year
* Normal mammogram within the last 13 months
* Normal Papanicolaou Test within the last 13 months

Exclusion Criteria:

* Serious intercurrent medical illnesses or history of seizure
* Significant cardiac disease (New York Heart Association Class III or IV)
* Abnormalities on the physical examination screen including significant abnormality of the heart, lungs, liver, spleen, or other abdominal organs, or neurologic abnormality Abnormalities on the biochemical screen that could be metabolically significant
* Individuals with intermediate equol values (> 10 ug/L to < 20 ug/L) on soy challenge
* Use of antibiotics within the last 3 months
* Use of hormone/estrogen therapy or SERMs within the last 3 months
* Abnormal thyroid or endocrine function tests; or current use of thyroid medication
* BMI at or above 35
* History of complete hysterectomy or oophorectomy
* High risk of breast cancer (5-year risk of >1.9%) based on NCI's Breast Cancer Risk Assessment Tool
* A history of a malignancy active or initially diagnosed within 2 years other than curatively treated non-melanoma carcinoma of the skin
* History of substance abuse or addiction
* Alcohol intake of greater than 2 drinks/day or 14 drinks/week
* Tobacco use
* Diets containing more than estimated intake of 20 mg genistein/day or 40mg isoflavone/day AND unwilling/unable to reduce soy intake to below this level during the study period
* Use of supplements containing phytoestrogens or that have estrogenic side effects within 1 month of study
* Pre-menopausal or pregnant
* Inability to read and comprehend the Informed Consent
* Life expectancy < 6 months
* History of breast cancer
* Known soy intolerance
* On chemotherapy within the last 2 years
* Inability to obtain an endometrial biopsy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-03; Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
DNA damage, apoptosis, estrogenic effects and changes in gene expression | 112 days

CONTACTS AND LOCATIONS:
Overall Officials: Steven H Zeisel, MD, PhD, Principal Investigator — UNC at Chapel Hill